CLINICAL TRIAL: NCT04281589
Title: Does End-Tidal Carbon Dioxide Value Show The Adequacy Of Ventilation In Low Tidal Volume Ventilation
Brief Title: End-tidal Carbon Dioxide Monitoring in Low Tidal Volume Ventilation
Acronym: ETCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: dondum
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Ventilation; End-Tidal Carbon Dioxide
Keywords: End-Tidal Carbon Dioxide; P(a-ET)CO2 gradient; ETCO2; low tidal volüm; mekanical Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: sequential
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): tidal volüm is 4 ml/kg
  Interventions: Other: if the ventilation parameter caused desaturation or hypercapnia we will change the parameter
- Group 2 (Experimental): tidal volüm is 6 ml/kg
  Interventions: Other: if the ventilation parameter caused desaturation or hypercapnia we will change the parameter
- Group 3 (Experimental): tidal volüm is 8 ml/kg
  Interventions: Other: if the ventilation parameter caused desaturation or hypercapnia we will change the parameter
- Group 4 (Experimental): tidal volüm is 10 ml/kg
  Interventions: Other: if the ventilation parameter caused desaturation or hypercapnia we will change the parameter

INTERVENTIONS:
Other: if the ventilation parameter caused desaturation or hypercapnia we will change the parameter — we will increased fi02

SUMMARY:
In cases where there is no ventilation-perfusion problem, the end-tidal carbon dioxide (ETCO2) value is closely associated with partial arterial carbon dioxide pressure (PaCO2); therefore, the PaCO2 value can be estimated using ETCO2 measurements in patients without significant cardiopulmonary disorders. The aim of the investigator's study is to evaluate the reliability of pulmonary ventilation monitoring with ETCO2 value and to investigate at what tidal volume values ETCO2 monitoring provides reliable information.

DETAILED DESCRIPTION:
The patients were grouped as follows: Group 1, if the tidal volume is 4 ml/kg; Group 2, if TV=6 ml/kg; Group 3, if TV=8 ml/kg; and Group 4, if TV=10 ml/kg. It was determined how many breaths per minute (minute ventilation) would be given with tidal volume x respiratory rate=6 L. The patients were ventilated with the same ventilation parameters for 30 minutes and then arterial blood gas analysis was performed. Arterial blood gas was collected at t1 for group 1, t2 for group 2, t3 for group 3, and t4 for group 4. The ETCO2 value, Peak pressure (Ppeak), Plateau pressure (Pplato), mean airway pressure (Pmean) values were recorded at the time of arterial blood gas collection. Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), peak heart rate (PHR) values were evaluated. The patients with a mean arterial pressure of less than 65 mmHg were excluded from the study. Partial arterial oxygen pressure (PaO2), partial arterial carbon dioxide pressure (PaCO2), oxygen saturation (SO2) values were recorded from the arterial blood gas analysis. P (a-ET) CO2 gradient value was calculated.

The groups were compared, in each patient, under the same conditions, when the different tidal volume was applied, how the ETCO2 monitorization, PaO2 values and hence the P (a-ET) CO2 gradient changed.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) classification 1, 2 risk group

Head and neck surgery under general anesthesia lasting more than 120 minutes and who progressed normotensive.

Exclusion Criteria:

Cardiac disease

Pulmonary disease

Obese patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
P (a-ET) CO2 gradient | 120 minutes
  The groups were compared, in each patient, under the same conditions, when the different tidal volume was applied, how the ETCO2 monitorization, PaCO2 values and hence the P (a-ET) CO2 gradient changed.

SECONDARY OUTCOMES:
Partial arterial oxygen pressure (PaO2) | 120 minutes
  Partial arterial oxygen pressure (PaO2) were recorded from the arterial blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Döndü Genç Moralar, Istanbul, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No